CLINICAL TRIAL: NCT02638532
Title: Volumetric Analysis in Autologous Fat Grafting to the Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jeffrey A. Gusenoff, MD, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15090106
Record Dates: First submitted 2015-12-11; First posted 2015-12-23 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Pedal Fat Pad Atrophy
Keywords: Fat Pad; Fat Pad Atrophy; Foot; Feet; Heel; Forefoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foot Fat Pad Grafting (Other): All subject who enter into the study will undergo the fat pad grafting procedure to either the Heel or Forefoot based on the discretion of the PI, Co-investigator and the study subject.
  Interventions: Procedure: Foot Fat Pad Grafting

INTERVENTIONS:
Procedure: Foot Fat Pad Grafting — Fat tissue to be used for grafting is harvested (usually from abdomen or thighs) with a small liposuction cannula. The fat tissue is then sterilely centrifuged and allowed to decant before separating the fluid and oil layers from the fat tissue fraction. The aspirated fat is then loaded into 1cc syringes and injected into the plantar fat pad using specialized injection cannulas.

SUMMARY:
The specific aim of this outcomes study is to assess if the volume of fat that is injected into the foot is retained at 6 months, to determine the retention over time, and assess the quality of the bone before and after treatment. We will also correlate adipose stem cell characteristics to the fat retention over time.

DETAILED DESCRIPTION:
The study goal is to utilize MRI to further understand changes that are occurring in the foot when autologous fat is used to treat plantar fat pad atrophy of the foot. The etiology of fat pad atrophy may be age-related, due to abnormal foot mechanics, obesity, steroid use, or collagen vascular disease. Displacement or atrophy of the fat pad can lead to osseous prominences in the foot that may be seen with painful skin lesions. Disease states, such as diabetes, may have loss of soft tissue integrity. Fat pad atrophy may result in significant pain or compensatory gait leading to callous formation or ulceration. In sensate patients, the pain can lead to emotional and physical pain, leading to productivity and financial losses.

Fat grafting to the feet is as a cosmetic surgery option. Although fat grafting is used often in standard care plastic surgery, for cosmetic reasons, it is considered part of the research in this trial. What happens to the fat after injection has not been well studied. Approximately 50 adults who experience pain from fat pad atrophy, either of the fore foot or heel will have fat pad grafting. The study will utilize MRI before and at 6 months post-procedure to assess changes in the quality of the bone of the foot as well as the 3D morphology of the fat. Specifically, the investigators want to know how the fat redistributes around the bone. In addition, the Adipose Stem Cell Biology Laboratory will assess the stem cell characteristics of the fat used for autotransplantation. This study will help build new collaborative efforts between Foot and Ankle Specialists, Stem Cell Biologists, and Plastic Surgeons, combining expertise in foot biomechanics with reconstructive fat grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, basically healthy and able to provide informed consent.
2. Patients with forefoot or rearfoot pain overlying the bone with fat pad atrophy.
3. At least 6 months post any surgical intervention to the foot.
4. Willing and able to comply with follow up examinations, including ultrasounds, MRI, and pedobarographic studies.
5. Diabetics: Type I and II with a HgA1C < or = 7.
6. Have tried and failed at least one form of conservative management (i.e. orthotics, padding, etc.).

Exclusion Criteria:

1. Age less than 18 years.
2. Inability to provide informed consent
3. Feet with open ulcerations or osteomyelitis.
4. Diabetics: Type I and II iwth a HgAIC > 7.
5. Active infection anywhere in the body.
6. Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment.
7. Known coagulopathy.
8. Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
9. Pregnancy.
10. Subjects with a diagnosis of Schizophrenia or Bipolar Disorder due to the inability to comply with study instructions, due in part to comorbidities (Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion).
11. Tobacco use: Last use within 1 year per patient report.
12. Patients with heart pacemakers, aneurysm clips, ear implants, IUD, shrapnel or metallic fragments in or on the body or eyes, neuro-stimulators, or other metal devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Utilize MRI to determine the 3D volumetric changes in the soft tissue of the foot after fat grafting and the changes in bone quality after fat grafting. | Baseline and 6 months post-procedure
  Comparative analysis of the scans will be done to note fat re-distribution and bone quality pre and post procedure.

SECONDARY OUTCOMES:
Ultrasound to measure tissue thickness of foot | Baseline, 1 month, 2 months and 6 months post-procedure
  Tissue thickness will be measured in MM. They will utilized to ascertain changes from pre procedure to 6 months post-procedure.
Pedobarograph to measure foot pressure and force while standing and walking | Baseline, 1 month, 2 months and 6 months post-procedure
  Foot pressure is measured in Kg/cm2 or psi. The pedobarograph provides imaging to show areas of distribution of pressure to the foot when subject stands and walks.
Adipose stem cell counts | Fat grafting procedure, 6 months
  excess fat from the procedure will be sent for stem cell analysis and used to corelate to retention of fat over time.
Manchester Foot Disability Index for pain | baseline, 1 month, 2 month and 6 month post procedure.
  Pain is assessed through the completion of a questionnaire that is scored.
Foot and Ankle Ability Measure for physical activity | baseline, 1 mont, 2 month, and 6 month post procedure.
  Activity level is assessed by subject rating different activities on the difficulty to complete the activities. The questionnaire is then scored.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery A Gusenoff, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Department of Plastic Surgery, Pittsburgh, Pennsylvania, United States